CLINICAL TRIAL: NCT02953782
Title: A Phase 1b/2 Trial of Hu5F9-G4 in Combination With Cetuximab in Patients With Solid Tumors and Advanced Colorectal Cancer
Brief Title: Study of Magrolimab (Hu5F9-G4) in Combination With Cetuximab in Participants With Solid Tumors and Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 5F9004
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Solid Tumor; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magrolimab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 (Experimental): Participants with solid tumor will receive a priming dose of magrolimab 1 mg/kg of body weight by intravenous (IV) infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 10 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 300 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 200 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, will start on Day 1. Each cycle will consist of 4 weeks (28 days). Cetuximab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented progressive disease (PD).
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with solid tumor will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 10 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, will start on Day 1. Each cycle will consist of 4 weeks (28 days). Cetuximab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with solid tumor will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 20 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, will start on Day 1. Each cycle will consist of 4 weeks (28 days). Cetuximab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with solid tumor will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, will start on Day 1. Each cycle will consist of 4 weeks (28 days). Cetuximab will be administered 1 hour prior to magrolimab infusion on days when both were given. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with solid tumor will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants will also receive a loading dose of magrolimab 45 mg/kg on Day 11 of Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab will start on Day 1 with weekly dose in Cycle 2 and bi-weekly dose in Cycle 3 onwards for magrolimab. Each cycle will consist of 4 weeks. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with advanced colorectal cancer (CRC) who are KRAS wild type (KRASwt) and are refractory to anti-EGFRmAb therapy will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab will start on Day 1; Days 8 and 22 are removed from Cycle 2 onwards for magrolimab. Each cycle will consist of 4 weeks. Cetuximab will be administered 1 hour prior to magrolimab infusion on days when both are given. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with advanced CRC with KRAS mutation (KRASm) who have progressed or are not candidates for oxaliplatin or irinotecan-based therapy will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab will start on Day 1; Days 8 and 22 are removed from Cycle 2 onwards for magrolimab. Each cycle will consist of 4 weeks. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab
- Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 (Experimental): Participants with advanced CRC with KRASm who have progressed or are not candidates for oxaliplatin or irinotecan-based therapy will receive a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approx. 3 hours) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approx. 2 hours) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants will also receive a loading dose of magrolimab 45 mg/kg of body weight on Day 11 of Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab will start on Day 1; Days 8 and 22 are removed from Cycle 3 onwards for magrolimab. Each cycle will consist of 4 weeks. Treatment will be administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
  Interventions: Drug: Magrolimab; Drug: Cetuximab

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: Hu5F9-G4
Drug: Cetuximab — Administered intravenously
  Other Names: ERBITUX®

SUMMARY:
The primary objectives of this study are: (Phase 1b) to investigate the safety and tolerability and to determine the recommended Phase 2 dose (RP2D) for magrolimab in combination with cetuximab; and (Phase 2) to evaluate overall response rate (ORR) of magrolimab in combination with cetuximab in participants with Kirsten rat sarcoma 2 viral oncogene homolog (KRAS) mutant and KRAS wild-type colorectal cancer (CRC).

ELIGIBILITY:
Key Inclusion Criteria:

* Histological Diagnosis

  * Phase 1b only: Advanced solid malignancy with an emphasis on colorectal cancer (CRC), head and neck, breast, pancreatic and ovarian cancers who have been treated with at least one regimen of prior systemic therapy, or who refuse systemic therapy, and for which there is no curative therapy available.
  * Phase 2:
* KRAS Mutant CRC: Advanced KRAS mutant CRC who have progressed or are ineligible for both irinotecan and oxaliplatin based chemotherapy
* KRAS Wild-Type CRC: Advanced KRAS wild type CRC who have progressed or are ineligible for fluoropyrimidine, irinotecan, and oxaliplatin based chemotherapy and who are relapsed or refractory to at least 1 prior systemic therapy that included an anti-epidermal growth factor receptor (EGFR) antibody, such as cetuximab, panitumumab or others.
* Adequate performance status and hematological, liver, and kidney function
* Phase 2 only: Willing to consent to 1 mandatory pre-treatment and 1 on-treatment tumor biopsy

Key Exclusion Criteria:

* Active brain metastases
* Prior treatment with cluster of differentiation 47 (CD47) or signal regulatory protein alpha (SIRPα) targeting agents.
* Phase 2 only: second malignancy within the last 3 years.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus (HIV)
* Pregnancy or active breastfeeding

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Wayne State University, Detroit, Michigan
  - START Midwest, Grand Rapids, Michigan
  - UPENN, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Md Anderson, Houston, Texas
  - START Center for Cancer Care, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 02 November 2016. The last study visit occurred on 10 February 2020.
Pre-assignment Details: 105 participants were screened.
Groups:
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by intravenous (IV) infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 10 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 300 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 200 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, started on Day 1. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented progressive disease (PD).
- Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 10 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, started on Day 1. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 20 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, started on Day 1. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, started on Day 1. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants also received a loading dose of magrolimab 45 mg/kg of body weight on Day 11 of Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1 with weekly dose in Cycle 2 and bi-weekly dose in Cycle 3 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced colorectal cancer (CRC) who were KRAS wild type (KRASwt) and were refractory to anti-EGFRmAb therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 2 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC with KRAS mutation (KRASm) who had progressed or were not candidates for oxaliplatin or irinotecan-based therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 2 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC with KRASm who had progressed or were not candidates for oxaliplatin or irinotecan-based therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants also received a loading dose of magrolimab 45 mg/kg of body weight on Day 11 of Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 3 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
Period: Phase 1b (Maximum Duration: 14.3 Months)
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Started | 6 | 3 | 9 | 8 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 3 | 9 | 8 | 6 | 0 | 0 | 0
Not completed — Death | 5 | 2 | 6 | 6 | 4 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Discontinued by Sponsor | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Participant placed in hospice care | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Period: Phase 2 (Maximum Duration: 11.1 Months)
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Started | 0 | 0 | 0 | 0 | 0 | 16 (11 participants were included in safety run-in to evaluate DLT. 9 out of 11 were evaluable for DLT.) | 15 | 15
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 16 | 15 | 15
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 14 | 11 | 8
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Not completed — Discontinued by Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Treated participants included all participants who received at least 1 dose of any study drugs.
Groups:
- Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 10 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 300 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 200 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1 and thereafter, weekly maintenance dose for both magrolimab and cetuximab, started on Day 1. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC who were KRASwt and were refractory to anti-EGFRmAb therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 2 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC with KRASm who had progressed or were not candidates for oxaliplatin or irinotecan-based therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 2 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Total: Total of all reporting groups
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Total
Number analyzed (Participants) | 6 | 3 | 9 | 8 | 6 | 16 | 15 | 15 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (6.72) | 68.6 (11.39) | 57.3 (7.05) | 52.4 (10.97) | 63.6 (9.50) | 59.7 (14.38) | 58.9 (14.41) | 57.4 (5.80) | 58.9 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 2 | 2 | 6 | 8 | 5 | 27
  Male | 4 | 3 | 7 | 6 | 4 | 10 | 7 | 10 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 8
  Not Hispanic or Latino | 5 | 3 | 8 | 8 | 5 | 12 | 13 | 11 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 5
  White | 5 | 3 | 7 | 8 | 6 | 8 | 10 | 8 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 4 | 3 | 4 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose Limiting Toxicities (DLT)
Description: DLT was defined as any Grade (GR) 3 or greater adverse event (AE) that was assessed as related to study treatment with the exceptions of:
  GR 3: anemia (hemolytic anemia that is medically significant tis considered a DLT), indirect/unconjugated hyperbilirubinemia, electrolyte abnormalities, elevation in alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase that resolved to ≤ Grade 2 with supportive care within 1 week and is not associated with other clinically significant consequences; nausea, vomiting, or diarrhea that resolved to ≤ Grade 2 with supportive care within 72 hours; fatigue that resolved to ≤ Grade 2 within 2 weeks on study; drug-related infusion reactions in the absence of an optimal pretreatment regimen; tumor lysis syndrome or electrolyte disturbances, hypomagnesemia, that resolved to ≤ Grade 2 or baseline within 1 week;
  GR 3 or 4: lymphopenia or leukopenia.
Time Frame: From first dose up to Day 28
Population: DLT Evaluable Analysis Set included participants who received at least 1 dose of any study drugs during Phase 1b if the participant either experienced a DLT any time during the DLT assessment period (the first 4 weeks of treatment) or completed at least 4 infusions of magrolimab and 2 infusions of cetuximab.
Measure: Number; unit: percentage of participants
Groups:
- Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2: Participants with solid tumor received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants also received a loading dose of magrolimab 45 mg/kg of body weight on Day 11 of Cycle 1.After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1 with weekly dose in Cycle 2 and bi-weekly dose in Cycle 3 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
- Phase 2 Cohort 1 Safety Run-in: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC who were KRASwt and were refractory to anti-EGFRmAb therapy received a maintenance dose of magrolimab 30 mg/kg of body weight by IV infusion (approximately 2 hours infusion) in combination with cetuximab 250 mg/m^2 infusions given over 60 minutes.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 Safety Run-in: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 6 | 3 | 9 | 7 | 6 | 9
percentage of participants | 16.7 | 0.0 | 0.0 | 14.3 | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE was any unfavorable and unintended sign, symptom, disease, and/or laboratory or physiological observation that may or may not be related to the investigational medicinal product. A TEAE was defined as AEs worsening or occurring during or after a participant's first exposure to study drug and within 30 days after the last administration of study drug or initiation of new anticancer therapy, whichever occurred first.
Time Frame: From first dose date up to last dose date plus 30 days (maximum: 15.3 months)
Population: All Treated included all participants who received at least 1 dose of any study drugs.
Measure: Number; unit: percentage of participants
Groups:
- Magrolimab Priming Dose Only: Participants who received only the priming dose (1 mg/kg) of magrolimab in Phase 2 of the study.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Magrolimab Priming Dose Only
Number analyzed (Participants) | 6 | 3 | 10 | 7 | 6 | 14 | 15 | 14 | 3
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

3. Primary Outcome: Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1)
Description: Objective response rate was defined as the percentage of participants with objective response which consisted of complete response (CR)+ partial response (PR) determined by RECIST v 1.1. CR: Disappearance of all target and all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (< 10 mm short axis). Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From Screening until 38.89 months (assessed on Day 1 of Cycle 3 then every 8 weeks [Q8W] from Cycle 5 onwards up to 38.89 months; 1 cycle = 4 weeks)
Population: Participants in All Treated with available data were analyzed. Efficacy results were planned to be reported separately for all CRC participants with KRASwt and KRASm tumors.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- KRASwt CRC: All CRC participants with KRASwt tumors who received assigned magrolimab doses in combination with cetuximab in any part of the study.
- KRASm CRC: All CRC participants with KRASm tumors who received assigned magrolimab doses in combination with cetuximab in any part of the study.
Arm/Group | KRASwt CRC | KRASm CRC
Number analyzed (Participants) | 32 | 42
percentage of participants | 6.3 [0.8 to 20.8] | 0.0 [0.0 to 8.4]

4. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Magrolimab
Description: Cmax is defined as the maximum concentration of drug.
Time Frame: Pre-magrolimab dose (within 12 hours) and 1-hour post-magrolimab dose (infusion duration = approximately 3 hours on Day 1 and 2 hours on other days) on Days 1 (Cycle 1 Day 1), 8 (Cycle 1 Day 8), and 29 (Cycle 2 Day 1) (1 cycle = 4 weeks)
Population: Participants in the PK Analysis Set (participants who received any amount of magrolimab with at least one detectable post-treatment serum concentration of magrolimab) with available data were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Groups:
- Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2: Participants with advanced CRC with KRAS mutation who had progressed or were not candidates for oxaliplatin or irinotecan-based therapy received a priming dose of magrolimab 1 mg/kg of body weight by IV infusion (approximately 3 hours infusion) on Day 1 followed by a maintenance dose of magrolimab 45 mg/kg of body weight by IV infusion (approximately 2 hours infusion) weekly starting on Day 8 followed by Days 15 and 22 in combination with cetuximab at a loading dose of 400 mg/m^2 infused over 120-minutes on Day 8 followed by a weekly maintenance dose of 250 mg/m^2 infusions given over 60 minutes on Days 15 and 22, in Cycle 1. Participants also received a loading dose of magrolimab 45 mg/kg of body weight on Day 11 of Cycle 1. After Cycle 1, maintenance dose for both magrolimab and cetuximab started on Day 1; Days 8 and 22 were removed from Cycle 3 onwards for magrolimab. Each cycle consisted of 4 weeks (28 days). Cetuximab was administered 1 hour prior to magrolimab infusion on days when both were given. Treatment was administered until unacceptable toxicity, voluntary withdrawal, or documented PD.
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 6 | 3 | 10 | 7 | 6 | 15 | 14 | 11
μg/mL
  Day 1 (Cycle 1 Day 1): number analyzed (Participants) | 6 | 2 | 10 | 7 | 6 | 15 | 11 | 11
  Day 1 (Cycle 1 Day 1) | 1.04 (0.769) | 0.629 (0.437) | 0.662 (0.374) | 0.432 (0.173) | 0.517 (0.311) | 0.479 (0.170) | 0.559 (0.254) | 0.525 (0.296)
  Day 8 (Cycle 1 Day 8): number analyzed (Participants) | 6 | 3 | 9 | 7 | 6 | 9 | 14 | 11
  Day 8 (Cycle 1 Day 8) | 209 (82.0) | 230 (54.6) | 455 (105) | 558 (168) | 1100 (287) | 513 (148) | 616 (121) | 901 (131)
  Day 29 (Cycle 2 Day 1): number analyzed (Participants) | 5 | 3 | 8 | 5 | 6 | 0 | 2 | 2
  Day 29 (Cycle 2 Day 1) | 312 (121) | 352 (68.4) | 728 (207) | 982 (182) | 2140 (590) |  | 775 (110) | 1790 (49.5)

5. Secondary Outcome: PK Parameter: Tmax of Magrolimab
Description: Tmax is defined as the time (observed time point) of Cmax.
Time Frame: Pre-magrolimab dose (within 12 hours) and 1-hour post-magrolimab dose (infusion duration = approximately 3 hours on Day 1 and 2 hours on other days) on Days 8 (Cycle 1 Day 8) and 29 (Cycle 2 Day 1) (1 cycle = 4 weeks)
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 6 | 3 | 9 | 7 | 6 | 9 | 14 | 11
days
  Day 8 (Cycle 1 Day 8) | 0.10 [0.09 to 0.12] | 0.12 [0.09 to 0.13] | 0.12 [0.12 to 6.94] | 0.14 [0.12 to 0.85] | 0.13 [0.12 to 3.90] | 0.12 [0.08 to 6.82] | 0.13 [0.12 to 0.17] | 0.12 [0.11 to 6.99]
  Day 29 (Cycle 2 Day 1): number analyzed (Participants) | 5 | 3 | 8 | 5 | 6 | 0 | 2 | 2
  Day 29 (Cycle 2 Day 1) | 0.94 [0.10 to 1.09] | 0.13 [0.12 to 0.13] | 0.13 [0.12 to 0.96] | 0.13 [0.10 to 0.15] | 0.12 [0.12 to 0.13] |  | 0.14 [0.14 to 0.14] | 0.12 [0.12 to 0.12]

6. Secondary Outcome: PK Parameter: AUClast of Magrolimab
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 5 | 3 | 9 | 6 | 6 | 1 | 0 | 0
day*μg/mL
  Day 8 (Cycle 1 Day 8): number analyzed (Participants) | 0 | 2 | 9 | 6 | 6 | 1 | 0 | 0
  Day 8 (Cycle 1 Day 8) |  | 676 (75.3) | 1530 (513) | 2140 (726) | 2920 (600) | 1930 |  |
  Day 29 (Cycle 2 Day 1): number analyzed (Participants) | 5 | 3 | 8 | 3 | 6 | 0 | 0 | 0
  Day 29 (Cycle 2 Day 1) | 1420 (711) | 1560 (413) | 3330 (1270) | 4480 (1220) | 7340 (2380) |  |  |

7. Secondary Outcome: PK Parameter: AUCtau of Magrolimab
Description: AUCtau is defined as concentration of drug over time (the area under the concentration verses time curve over the dosing interval).
Time Frame: as for outcome 5
Population: Participants in the PK Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: day*μg/mL
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 6 | 4 | 1 | 0 | 0
day*μg/mL
  Day 8 (Cycle 1 Day 8): number analyzed (Participants) | 0 | 2 | 5 | 6 | 0 | 1 | 0 | 0
  Day 8 (Cycle 1 Day 8) |  | 676 (75.3) | 1630 (649) | 2140 (726) |  | 1930 |  |
  Day 29 (Cycle 2 Day 1): number analyzed (Participants) | 4 | 3 | 7 | 3 | 4 | 0 | 0 | 0
  Day 29 (Cycle 2 Day 1) | 1640 (604) | 1560 (413) | 3630 (1040) | 4480 (1220) | 8770 (1120) |  |  |

8. Secondary Outcome: Percentage of Participants With Anti-drug Antibodies (ADA)
Description: Percentage of Participants With Positive ADA at any timepoint was reported.
Time Frame: Baseline; post-treatment (assessed continuously up to 30 days after last dose; maximum 15.3 months )
Population: Immunogenicity Analysis Set included participants with at least one reported ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b Cohort 1: Magrolimab 10 mg/kg + Cetuximab 200 mg/m^2 | Phase 1b Cohort 2: Magrolimab 10 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 3: Magrolimab 20 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 4: Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 1b Cohort 5: Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 1 (KRASwt): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 2 (KRASm): Magrolimab 30 mg/kg + Cetuximab 250 mg/m^2 | Phase 2 Cohort 3 (KRASm): Magrolimab 45 mg/kg + Cetuximab 250 mg/m^2
Number analyzed (Participants) | 6 | 3 | 10 | 7 | 6 | 16 | 15 | 15
percentage of participants
  Baseline ADA | 0.00 | 0.00 | 0.00 | 14.3 | 0.00 | 6.3 | 0.00 | 0.00
  Post-Treatment ADA: number analyzed (Participants) | 6 | 3 | 10 | 7 | 6 | 16 | 15 | 14
  Post-Treatment ADA | 33.3 | 0.00 | 0.00 | 0.00 | 0.00 | 6.3 | 13.3 | 0.00
  Overall ADA | 33.3 | 0.00 | 0.00 | 14.3 | 0.00 | 12.5 | 13.3 | 0.00

9. Secondary Outcome: Disease Control Rate (DCR) as Assessed by RECIST v1.1
Description: DCR was defined as the percentage of participants with disease control which consisted of CR+PR+SD. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters measured while on study. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions.
Time Frame: From Screening until 38.89 months (assessed on Cycle 3 Day 1 then every 8 weeks from Cycle 5 onwards up to 38.89 months; 1 cycle = 4 weeks)
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | KRASwt CRC | KRASm CRC
Number analyzed (Participants) | 32 | 42
percentage of participants | 50.0 [31.9 to 68.1] | 38.1 [23.6 to 54.4]

10. Secondary Outcome: Duration of Response (DOR) as Assessed by RECIST v1.1
Description: DOR was measured from when the first (objective) response was met (i.e., CR or PR) until the first date of objectively documented PD. Participants who did not have objectively PD was censored at their last documented progression-free date. CR: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) had a reduction in short axis to < 10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Kaplan Meier estimate was used for analysis.
Time Frame: From first objective response until documented PD (assessed on Cycle 3 Day 1 then every 8 weeks from Cycle 5 onwards up to 38.89 months; 1 cycle = 4 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRASwt CRC | KRASm CRC
Number analyzed (Participants) | 2 | 0
months | 9.7 [7.0 to 12.5] |

11. Secondary Outcome: Progression Free Survival (PFS) as Assessed by RECIST v1.1
Description: PFS was measured from first dose until the first date of objectively documented PD or death. Participants who did not have objectively documented PD and not died was censored at their last documented progression-free date. PD: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum measured while on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Unequivocal progression of existing non-target lesions. Kaplan Meier estimate was used for analysis.
Time Frame: From first dose until documented PD/death (assessed on Cycle 3 Day 1 then every 8 weeks from Cycle 5 onwards up to 38.89 months; 1 cycle = 4 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRASwt CRC | KRASm CRC
Number analyzed (Participants) | 32 | 42
months | 3.6 [1.8 to 5.4] | 1.9 [1.8 to 3.5]

12. Secondary Outcome: Overall Survival (OS)
Description: OS was measured from first dose until death. Participants who did not die were censored at their last known alive date. Kaplan Meier estimate was used for analysis.
Time Frame: From first dose until death (assessed on Cycle 3 Day 1 then every 8 weeks from Cycle 5 onwards up to 38.89 months; 1 cycle = 4 weeks)
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | KRASwt CRC | KRASm CRC
Number analyzed (Participants) | 32 | 42
months | 9.5 [5.9 to 12.6] | 7.6 [5.4 to 11.7]

ADVERSE EVENTS:
Time Frame: Adverse Events: From first dose date up to last dose date plus 30 days (maximum: 15.3 months); All-Cause mortality: From first dose date up to 38.89 months
Description: All Treated participants included all participants who received at least 1 dose of any study drugs. Per planned analysis, AE data were summarized by the magrolimab maintenance dose level.
Groups:
- Magrolimab 10 mg/kg: Participants who received magrolimab maintenance dose of 10 mg/kg in combination with cetuximab in any part of the study.
- Magrolimab 20 mg/kg: Participants who received magrolimab maintenance dose of 20 mg/kg in combination with cetuximab in any part of the study.
- Magrolimab 30 mg/kg: Participants who received magrolimab maintenance dose of 30 mg/kg in combination with cetuximab in any part of the study.
- Magrolimab 45 mg/kg: Participants who received magrolimab maintenance dose of 45 mg/kg in combination with cetuximab in any part of the study.
Arm/Group | Magrolimab 10 mg/kg | Magrolimab 20 mg/kg | Magrolimab 30 mg/kg | Magrolimab 45 mg/kg | Magrolimab Priming Dose Only
All-Cause Mortality (participants affected / at risk) | 7/9 | 8/10 | 30/36 | 14/20 | 3/3
Serious Adverse Events (participants affected / at risk) | 3/9 | 6/10 | 10/36 | 5/20 | 1/3
Other Adverse Events (participants affected / at risk) | 9/9 | 10/10 | 36/36 | 20/20 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab 10 mg/kg (N=9) | Magrolimab 20 mg/kg (N=10) | Magrolimab 30 mg/kg (N=36) | Magrolimab 45 mg/kg (N=20) | Magrolimab Priming Dose Only (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 1 | 1 | 0
Complication associated with device (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 3 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab 10 mg/kg (N=9) | Magrolimab 20 mg/kg (N=10) | Magrolimab 30 mg/kg (N=36) | Magrolimab 45 mg/kg (N=20) | Magrolimab Priming Dose Only (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 11 | 4 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 1 | 0 | 0
Blepharal pigmentation (Eye disorders) | 0 | 0 | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 1 | 0 | 0
Photopsia (Eye disorders) | 1 | 2 | 2 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 3 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 3 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 3 | 4 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3 | 6 | 2 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 5 | 6 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 9 | 7 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Loose tooth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 16 | 3 | 1
Oesophageal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rectal discharge (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 8 | 6 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 11 | 4 | 1
Chest discomfort (General disorders) | 1 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 2 | 11 | 5 | 0
Early satiety (General disorders) | 0 | 1 | 1 | 1 | 0
Fatigue (General disorders) | 4 | 5 | 18 | 7 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 3 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 2 | 0 | 2 | 2 | 0
Pain (General disorders) | 0 | 0 | 3 | 0 | 1
Performance status decreased (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 2 | 13 | 8 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Nail infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Tinea cruris (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 1 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 12 | 7 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 2 | 4 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 2 | 5 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 2 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 3 | 5 | 5 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 4 | 1 | 3 | 3 | 0
Platelet count decreased (Investigations) | 1 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 3 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 9 | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 4 | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 5 | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 10 | 5 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 5 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 2 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 2 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 17 | 8 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 0 | 4 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 3 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 2 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 4 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 11 | 3 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 5 | 14 | 6 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 3 | 8 | 10 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 7 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 7 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 3 | 7 | 5 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 2 | 1 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT02953782/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-12): https://cdn.clinicaltrials.gov/large-docs/82/NCT02953782/SAP_001.pdf